CLINICAL TRIAL: NCT03366207
Title: Clinical and Microbiologic Efficacy of Ciprofloxacin for the Treatment of Uncomplicated Urinary Tract Infection in Adult Women.
Brief Title: Efficacy of Ciprofloxacin for the Treatment of Uncomplicated Urinary Tract Infection (uUTI)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Iterum Therapeutics, International Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IT004-401
Record Dates: First submitted 2017-12-04; First posted 2017-12-08 (Actual); Results first posted 2019-08-21 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-07

CONDITIONS: UTI - Lower Urinary Tract Infection; Antibiotic Resistant Infection
MeSH Terms: interventions — Ciprofloxacin

STUDY DESIGN:
Intervention Model Description: Open label study of ciprofloxacin for uncomplicated urinary tract infection
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Ciprofloxacin (Experimental): Ciprofloxacin for the treatment of uncomplicated urinary tract infection
  Interventions: Drug: Ciprofloxacin

INTERVENTIONS:
Drug: Ciprofloxacin — Ciprofloxacin 250 mg PO twice daily (BID) x 3 days for women with uUTI.
  Other Names: Cipro

SUMMARY:
This is a prospective, Phase 4, open label, multi-center study of the clinical and microbiologic efficacy of ciprofloxacin for the treatment of uncomplicated urinary tract infections in adult women.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients ≥18 years of age with more than 24 hours of urinary symptoms attributable to a UTI
2. Two of the following signs and symptoms of uUTI: urinary frequency, urinary urgency, pain or burning on micturition, suprapubic pain, gross hematuria
3. A mid-stream urine specimen with:

   1. a dipstick analysis positive for nitrite AND
   2. a dipstick analysis positive for leukocyte esterase
4. Has given written informed consent to participate in the study.

Exclusion Criteria:

1. Presence of signs and symptoms suggestive of acute pyelonephritis: fever (temperature > 38°Celsius), chills, costovertebral angle tenderness, flank pain, nausea and/or vomiting
2. Receipt of prior effective antibacterial drug therapy for uUTI for the presenting illness unless the recovered pathogen demonstrates resistance to initial antibiotic and clinical symptoms persist
3. Concurrent use of non-study antibacterial drug therapy that would have a potential effect on outcome evaluations in patients with uUTI
4. Patients with ileal loops or urinary stoma
5. Patients with an indwelling urinary catheter in the previous 30 days
6. Patients with paraplegia
7. Patients who are likely to receive ongoing antibacterial drug prophylaxis after treatment of uUTI (e.g., patients with vesico-ureteral reflux)
8. Any history of trauma to the pelvis or urinary tract
9. Patient's urine culture results, if available at study entry, identify more than 2 microorganisms regardless of colony count or patient has a potential fungal pathogen
10. Patient's urine culture results, if available at study entry, identifies the causative uropathogen for the presenting illness to be resistant to ciprofloxacin
11. Patient has severe chronic kidney disease, or is receiving hemodialysis or peritoneal dialysis or had a renal transplant
12. Patient is known to have severe neutropenia
13. Patient is known to be pregnant
14. Patients with uncontrolled diabetes mellitus
15. Patients with a known history of myasthenia gravis
16. Patients who require concomitant administration of tizanidine
17. Patients with a history of allergy to quinolones
18. Patient is considered unlikely to survive the study period or has a rapidly progressive or terminal illness including septic shock which is associated with a high risk of mortality

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only females are eligible to participate in this study.
Enrollment: 250 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Aronin, MD, Principal Investigator — Iterum Therapeutics
Locations (1):
- Restore Clinical Research, Cary, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ciprofloxacin
Started | 250
Completed | 242
Not Completed | 8

BASELINE CHARACTERISTICS:
Arm/Group | Ciprofloxacin
Number analyzed (Participants) | 250
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 205
  >=65 years | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.3 (16.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 250
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 147
  Not Hispanic or Latino | 98
  Unknown or Not Reported | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 42
  White | 202
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 250
Body-mass index [Mean (Standard Deviation); unit: kg/m^2] | 29.01 (6.861)

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Combined Clinical and Microbiologic Response
Description: Clinical response is defined as complete resolution of uUTI symptoms at entry and no new uUTI symptoms; microbiologic success is defined as eradication of baseline pathogen
Time Frame: From start of treatment until assessment of cure, approximately 12 days
Population: Microbiological modified intent to treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Ciprofloxacin
Number analyzed (Participants) | 124
Participants | 70

2. Secondary Outcome: Microbiologic Response
Description: Microbiologic response is defined as demonstrating <1000 colony-forming units per mL of the baseline uropathogen at the test of cure visit
Time Frame: From start of treatment until assessment of cure, approximately 12 days
Population: Microbiological modified intent to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Ciprofloxacin
Number analyzed (Participants) | 124
Participants | 96

ADVERSE EVENTS:
Time Frame: From start of treatment until assessment of cure, approximately 12 days
Arm/Group | Ciprofloxacin
All-Cause Mortality (participants affected / at risk) | 0/242
Serious Adverse Events (participants affected / at risk) | 0/242
Other Adverse Events (participants affected / at risk) | 0/242

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator may publish/present results provided the following are satisfied: (i) Sponsor consents to publication; (ii) Multi-Center Publication published; or at least 18 months since database lock; (iii) investigator must submit proposed publication to Sponsor for review, allowing at least 60 days to review. The Investigator shall delay publication/presentation for up to 45 days to permit the Sponsor time to obtain Intellectual Property protections and protect confidential information.

DOCUMENTS (2):
  • Study Protocol (2018-03-27): https://cdn.clinicaltrials.gov/large-docs/07/NCT03366207/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-30): https://cdn.clinicaltrials.gov/large-docs/07/NCT03366207/SAP_001.pdf